CLINICAL TRIAL: NCT06832358
Title: Effect Evaluation of PERMA Positive Psychological Intervention Model in Parkinson's Disease Patients
Brief Title: Positive Psychological Intervention for Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Meichun Shu, Doctor, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Meichun Shu2
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Parkinson

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): The study group was treated with routine nursing combined with PERMA positive psychological intervention mode
  Interventions: Behavioral: Routine nursing methods; Behavioral: PERMA positive psychological intervention mode
- Control group (Active Comparator): The control group will receive routine nursing methods to ensure that patients receive standard medical support and treatment during the intervention period.
  Interventions: Behavioral: Routine nursing methods

INTERVENTIONS:
Behavioral: Routine nursing methods — According to their condition, they receive individualized drug treatment, including the main drugs of Parkinson's disease (such as dopamine replacement drugs) and combined antidepressant drugs. Secondly, regular follow-up evaluations will be conducted to monitor disease progression and drug side effects. At the same time, patients and their families will receive health education on Parkinson's disease and depression.The patients would receive basic psychological support. Medical staff will encourage patients to express their emotions and pay attention to their psychological state, which will help alleviate anxiety and depression. Medical staff will provide patients with information about local support organizations and social groups, and encourage patients to participate in related activities to increase social interaction and emotional support.
Behavioral: PERMA positive psychological intervention mode — (1) Formation of an intervention team.(2) Development and execution of interventions.The study group participated in a series of positive psychology workshop involving interviews and exercises aligned with the PERMA model as part of their routine health education. Each participant took part in individualized interviews focused on two specific topics each week until all subjects were covered, with each session lasting between 30 to 50 minutes. This interview phase continued for one month, conducted in the hospital ward.
  Arms: Study group

SUMMARY:
This study aims to evaluate the impact of positive psychological intervention based on the PERMA model on Parkinson's disease patients by assessing their depression, quality of life, and related psychological indicators before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the clinical diagnostic criteria for primary Parkinson's disease
* Subjects must not have a history of depression or other significant illnesses (e.g., stroke, coronary heart and tumor disease)
* Subjects should have clear consciousness, effective communication capabilities, and basic comprehension and reading skills to complete routine assessments
* The diagnosis of depression adhered to the ' Chinese Classification and Diagnostic Criteria for Mental Disorders ' (Revised Third Edition)
* Subjectsshould not have schizophrenia
* Subjects should not have substance abuse (alcohol, tobacco or other psychoactive substances)

Exclusion Criteria:

* Subjects with significant mental or cognitive impairment that communication or completion of scale assessments
* Subjects exhibiting severe self-harm or suicidal tendencies
* Subjects with severe dysfunction of the heart, liver, kidney or other critical organs
* Subjects with contraindications for transcranial magnetic stimulation (such as cochlear implant, pacemaker, built-in pump, artificial metal heart valve, suspected metal in the eye or elevated intracranial pressure)
* Subjects with a history of epilepsy that is poorly controlled
* Subjects with Parkinson's disease who have undergone surgical treatment

Ages: 42 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
the scores of Unified Parkinson's Disease Rating Scale(UPDRS) | before the intervention
the scores of Unified Parkinson's Disease Rating Scale(UPDRS) | after one month of intervention
the scores of Parkinson's Disease Quality of Life Scale(PDQ-39) | before the intervention
the scores of Parkinson's Disease Quality of Life Scale(PDQ-39) | after one month of intervention
the scores of Hamilton Depression Scale(HAMD) | before the intervention
the scores of Hamilton Depression Scale(HAMD) | after one month of intervention
the scores of Hamilton Anxiety Scale(HAMA) | before the intervention
the scores of Hamilton Anxiety Scale(HAMA) | after one month of intervention
the scores of Connor-Davidson Resilience Scale(CD-RISC) | before the intervention
the scores of Connor-Davidson Resilience Scale(CD-RISC) | after one month of intervention
the scores of Pittsburgh Sleep Quality Index(PSQI) | before the intervention
the scores of Pittsburgh Sleep Quality Index(PSQI) | after one month of intervention
the scores of Mini-Mental State Examination(MMSE) | before the intervention
the scores of Mini-Mental State Examination(MMSE) | after one month of intervention
the scores of Positive and Negative Affect Schedule (PANAS) | before the intervention
the scores of Positive and Negative Affect Schedule (PANAS) | after one month of intervention
the Newcastle Nursing Satisfaction Scale score | before the intervention
the Newcastle Nursing Satisfaction Scale score | after one month of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, China

IPD SHARING:
Plan to Share IPD: Undecided